CLINICAL TRIAL: NCT06975631
Title: Post-market Study for the Evaluation of the Effectiveness and Safety of Treatment With TrHCROSS by i+Med in Knee Osteoarthritis After a Single Intra-articular Administration
Brief Title: Post-market Study on TrHCROSS® in Knee Osteoarthritis After a Single Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Hospital Universitario Araba (Other); Bioaraba (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TrHCROSS-PIC01-2021
Record Dates: First submitted 2025-04-23; First posted 2025-05-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
Keywords: KOA; Osteoarthritis; Knee; Sodium Hyaluronate; WOMAC; VAS; KOOS
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Non-inferiority, controlled, interventional, randomized, parallel-group, single-blind, and single-center clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TrHCROSS® (Experimental): Class II medical device based on a sterile viscoelastic solution of cross-linked sodium hyaluronate, indicated as an intra-articular viscoelastic supplement for the treatment of osteoarthritis symptoms
  Interventions: Device: TrHCROSS®
- Hyalone® (Active Comparator): Class II medical device based on a sterile sodium hyaluronate solution that restores the viscoelastic properties of synovial fluid, relieving pain and improving mobility in degenerative joint disorders
  Interventions: Device: Hyalone®

INTERVENTIONS:
Device: TrHCROSS® — Single injection of 4.4 ml of viscoelastic sodium hyaluronate solution crosslinked.
  Arms: TrHCROSS®
Device: Hyalone® — Single injection of 4.4 ml of viscoelastic sodium hyaluronate solution crosslinked
  Arms: Hyalone®

SUMMARY:
Double-blind study assessing the safety and efficacy of TrHCROSS® in knee osteoarthritis, compared to Hyalone®, using scales such as WOMAC, VAS, and KOOS. The population includes 60 symptomatic patients with mild to moderate KOA (Kellgren-Lawrence II or III) who have not responded adequately to non-pharmacological treatments or simple analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 80 years of age.
* Body mass index <40 kg/m².
* Diagnosis of knee osteoarthritis (KOA). The stage must be radiographically confirmed (Kellgren-Lawrence grade II or III) within 6 months prior to study entry.
* Persistent pain reported during the 3 months prior to recruitment and moderate to severe pain when walking on inclines or stairs, or at rest (VAS score ≥40) at baseline.
* History of analgesic use (paracetamol and/or NSAIDs) related to the study condition.
* Willingness and ability to complete questionnaires and understand study instructions.
* Signed informed consent specific to the study.

Exclusion Criteria:

* X-rays showing grade IV changes on the Kellgren-Lawrence scale.
* Severe functional impairment in the knee.
* Bilateral involvement (simultaneous involvement of both knees).
* Associated hip osteoarthritis.
* Clinically significant pain in joints other than the knee.
* Psoriasis.
* Patients with confirmed rheumatic joint disease.
* Active infection.
* Known or suspected use of intra-articular steroids within the previous 3 months, or intra-articular HA or PRP within the 9 months prior to treatment initiation, as well as the use of chondroprotective agents.
* Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of TrHCROSS® for pain relief in patients with KOA. | In 24 weeks.
  Comparison of TrHCROSS® with Hyalone®, with significant improvement considered if there was a change of ≥50% and ≥5 points in the WOMAC A pain score.
  The WOMAC A questionnaire is divided into five items to measure pain, with a scoring range from 0 to 20, where 0 represents the least amount of pain and 20 represents the most intense pain.
Serious adverse events. | Through study completion, approximately 52 weeks.
  Evaluate the safety of the treatment, in terms of the incidence of serious adverse events.

SECONDARY OUTCOMES:
Pain relief using WOMAC A. | At the conclusion of the study, approximately 52 weeks later.
  Evaluate the effectiveness of TrHCROSS® in pain relief at 52 weeks using the WOMAC A pain score, and compare it with Hyalone®. The WOMAC A questionnaire consists of five items to assess pain, with a scoring range from 0 to 20, where 0 indicates minimal pain and 20 represents the most severe pain.
Stiffness using WOMAC B. | In 24 weeks and in 52 weeks.
  Assess the effectiveness of TrHCROSS® in reducing stiffness at 24 and 52 weeks using the WOMAC B stiffness score, and compare it with Hyalone®. The WOMAC B questionnaire ranges from 0 to 8, where a lower score reflects less stiffness and a higher score indicates more severe stiffness.
Functionality using WOMAC C. | In 24 weeks and in 52 weeks.
  Evaluate the effectiveness of TrHCROSS® in improving functionality at 24 and 52 weeks using the WOMAC C functionality score, and compare it with Hyalone®. The WOMAC C questionnaire has a scoring range from 0 to 68, where a lower score indicates less difficulty and a higher score indicates greater difficulty.
Global Patient Assessment. | In 24 weeks and in 52 weeks.
  Analyze the global patient assessment after administration of the study treatment with VAS and compare it with the one obtained after administration of Hyalone®.
  The Visual Analogue Scale (VAS) allows for the assessment of the patient's overall evaluation, ranging from 0 to 100 mm, with 0 indicating the best outcome and 100 the worst outcome.
Combined WOMAC and VAS scales. | At baseline, in 24 weeks and in 52 weeks.
  Evaluate the combined WOMAC and VAS scales from baseline at all follow-up visits (weeks 24 and 52). The VAS is measured in mm (from 0 to 100), while the WOMAC uses a Likert scale to provide a total score.
Improvement in pain score. | At baseline, in 24 weeks and in 52 weeks.
  Analyze the improvement in pain scores (WOMAC A) from baseline (at least 40% and ≥5 points) in each treatment group separately. The WOMAC A questionnaire consists of five items to assess pain, with a scoring range from 0 to 20, where 0 indicates minimal pain and 20 represents the most severe pain.
Improvement in KOOS scores. | At baseline, in 24 weeks and in 52 weeks.
  Analyze the significant improvement in KOOS scores from baseline in each treatment group separately.
  The KOOS scale is divided into subscales that are scored individually: Pain, Other Symptoms, Daily Activities, Function, Sports/Recreational Activities, and Quality of Life. A Likert scale is used, and all items have five possible options ranging from 0 (No problems) to 4 (Extreme problems). Each of the five scores is calculated as the sum of the items included
Treatment response rate. | At baseline, in 24 weeks and in 52 weeks.
  Calculate the treatment response rate at all follow-up visits (weeks 24 and 52) according to the OMERACT-OARSI criteria and compare it with Hyalone®. A responder is defined as having at least a 50% improvement and an absolute change of ≥20mm in pain or functionality, or improvement in two of the three subscales with ≥20% and ≥10mm change in the VAS scales for pain, functionality, and overall patient evaluation.
Patient satisfaction with treatment. | At the conclusion of the study, approximately 52 weeks later.
  Evaluate patient satisfaction with the treatment using a Likert scale with 5 options: Very satisfied, Satisfied, Slightly satisfied, Indifferent, and Dissatisfied. The percentage of patients who rate their satisfaction as 'Very satisfied,' 'Satisfied,' and 'Slightly satisfied' will be calculated.
Other adverse events. | Through study completion, approximately 52 weeks.
  Analyze and record the incidence of other adverse events to ensure it does not exceed the pre-established threshold of 18%.
Analgesic use. | Through study completion, approximately 52 weeks.
  Monitor the need for analgesic use.
Joint mobility. | At baseline, in 24 weeks and in 52 weeks.
  Evaluate joint mobility by measuring the joint range with a goniometer and assess its progression from baseline to the follow-up visits.
Investigator´s global assessment. | At the conclusion of the study, approximately 52 weeks later.
  For the overall treatment evaluation by the investigator, a Likert scale with 5 options will be used: Significant improvement, Improvement, Slight improvement, No change, and Worsening. Patients classified by the investigator as having a perceived global change after treatment of 'slight improvement,' 'improvement,' or 'significant improvement' will be identified as having a clinically relevant improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Álava, Vitoria-Gasteiz, Álava, Spain